CLINICAL TRIAL: NCT02844218
Title: Effect of Age on Treatment Decision-Making in Elderly Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0463
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Chemotherapy; Low-intensity therapy; Older patients; Prognosis; Supportive care
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Intensive chemotherapy group: Group 1: Patients' age ≥ 70 years treated from 1985 to 1999 with intensive induction chemotherapy.
  Interventions: Other: Age of patient
- Lower intensity treatment group: Group 2: patients treated from 2000 to 2006 with intensive chemotherapy plus improved supportive care and a follow-up protocol systematically performed at the university hospital.
  Interventions: Other: Age of patient
- personalized treatment group: Group 3: patients who had received, starting in 2007, more "personalized" treatment with either intensive chemotherapy or lower-intensity therapy determined by the clinical judgment of the treating physician.
  Interventions: Other: Age of patient

INTERVENTIONS:
Other: Age of patient — * Historical Comparison Between Patients Aged 60 to 69 and Patients Aged ≥ 70 Years Treated With Intensive Chemotherapy.
  * Comparison between Intensive Chemotherapy and Low-Intensity Treatments in Patients Aged ≥70 Years.
  * Improvement of Treatments Over Time
  * Overall Survival (OS) of patients aged ≥ 70 Years during3 study periods. Period 1, from 1985 to 1999, during which all patients with acute Myeloid Leukemia received an intensive chemotherapy regimen at the University Hospital. Period 2, from 2000 to 2006, during which all patients received an Intensive Chemotherapy regimen, Improved Supportive Care and follow-Up protocol at the University Hospital. Period 3, From 2007 to 2014, during Which patients received Improved Supportive Care and follow-up protocol at the University Hospital and "Personalized" Therapy (Intensive Chemotherapy or Low-Dose Intensity Treatment)

SUMMARY:
Patients aged ≥70 years with acute myeloid leukemia (AML) have a poorer prognosis than those aged 60 to 69 years. The poor outcome is the result of treatment-related toxicity in elderly patients, owing to comorbidities, the greater possibility of other hematopoietic disorders, and a biologically poor risk prognosis. Anthracycline- and cytarabine-based therapy, administered for 3 and 7 days respectively (3 +7), remains the standard induction therapy for this patient population. This approach improved survival compared with supportive care (median, 5 vs. 3 months) for adults aged ≥ 65 years. However, the overall view has been that the results of intensive chemotherapy in elderly patients remain poor. Although complete remission (CR) rates of 40% to 80% can be achieved in highly selected populations, long-term survival has been poor. Furthermore, most clinical trials have only enrolled patients with an adequate performance status (PS).

Prognostic models have been developed from clinical trial data to predict the outcomes for older patients. However; each model relies on chronologic age. Age is a surrogate measure for both changes in tumor biology and patient characteristics. Understanding which patients are likely to benefit from intensive therapies versus low-intensity therapies or supportive care is critical. The definition of "fit" to undergo intensive induction therapy has not been established, and the therapeutic choice is mainly determined by physician and patient decision. In older patients, low-dose cytarabine (LD-AraC) has been demonstrated to be more beneficial than best supportive care and hydroxyurea. The recent availability of new drugs that could have an improved side effect profile and, in some cases, bioavailability might offer future improvement for this patient population. In this setting, the investigators have tended to consider, since 2007, patients aged ≥70 years as potential candidates for alternative lower intensity therapy (LD-AraC, hypomethylating agents) even when they presented in good physical condition.

The investigators goal was to determine whether age ≥ 70 years could represent a useful and simple cut off for treatment decision-making in clinical practice and whether low-intensity therapy could be an alternative therapeutic approach to intensive chemotherapy even for patients aged ≥ 70 years who were theoretically "fit" (WHO /ECOG/ PS of ≤ 2).

ELIGIBILITY:
Inclusion Criteria:

* Are at least 70 years of age
* Have a diagnosis of AML according to World Health Organization (WHO) classification
* Provide signed, written informed consent

Exclusion Criteria:

* Patients with acute promyelocytic leukemia
* Have an ECOG score ≥2

Ages: 70 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Acute myeloid leukemia (AML)
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Date of last contact if alive (up to 11 months)
  OS was the main endpoint for this analysis. The event for OS was death, and patients were censored at the date of last contact, if alive.

SECONDARY OUTCOMES:
Complete remission rate (CR) | Date of last contact if alive or death (up to 11 months)
  A CR was defined according to standard criteria as < 5% blasts in bone marrow aspirates with evidence of maturation of cell lines and restoration of the peripheral blood counts.
First Relapse | Duration of the study (11 months)
  Hematologic relapse was considered when > 5% blasts were seen in 2 bone marrow aspirates obtained at a 15-day interval.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier THOMAS, MD-PhD, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud
Locations (1):
- Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, 165 Chemin du Grand Revoyet, Pierre-Bénite, France